CLINICAL TRIAL: NCT02827799
Title: Cognitive Behavioral Therapy for Insomnia in Stable Heart Failure
Acronym: CBTI-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 0904005041_B; R21NR011387 (NIH)
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Heart Failure; Insomnia; Cardiomyopathy
Keywords: heart failure; insomnia; sleep disorders; actigraphy; cardiomyopathy; depression; sleepiness; anxiety; fatigue
MeSH Terms: conditions — Heart Failure; Sleep Initiation and Maintenance Disorders; Cardiomyopathies; Sleep Wake Disorders; Depression; Sleepiness; Anxiety Disorders; Fatigue | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heart Failure Self-Management Education (Placebo Comparator): This treatment includes participation in 4 one hour biweekly face-face sessions of education on heart failure self-management, as well as a 15 minute telephone call on intervening weeks. The total intervention is 8 weeks.
  Interventions: Behavioral: Heart Failure Self-Management Education
- Cognitive Behavioral Therapy for Insomnia (CBT-I) (Experimental): This treatment includes participation in 4 one hour biweekly face-face sessions of cognitive behavioral therapy for insomnia, as well as a 15 minute telephone call on intervening weeks. The total intervention is 8 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — This behavioral intervention includes training on managing the sleep environment (stimulus control), managing dysfunctional beliefs and attitudes about sleep (cognitive therapy), relaxation (progressive muscle relaxation), changing sleep behaviors (sleep hygiene), and managing sleep duration and continuity (sleep restriction).
  Arms: Cognitive Behavioral Therapy for Insomnia (CBT-I)
Behavioral: Heart Failure Self-Management Education — This intervention includes learning about how to manage one's heart failure. This includes understanding when to seek treatment, monitoring oneself for daily signs and symptoms, daily weight, dietary changes, physical activity, and adherence to medication taking.
  Arms: Heart Failure Self-Management Education

SUMMARY:
The purpose of this exploratory developmental study is to test the feasibility, acceptability, and preliminary efficacy of cognitive behavioral therapy for insomnia (CBT-I) among adults who have stable Heart Failure. Participants were randomized either to a treatment (CBT-I) or attention-control condition (heart failure self management education).

DETAILED DESCRIPTION:
Insomnia is common in adults with chronic heart failure (HF), a condition associated with functional performance deficits, symptom burden, and high levels of morbidity and mortality. To date there has been little study of strategies to improve sleep in this large population. Cognitive behavioral therapy for insomnia (CBT-I) is an effective treatment for insomnia comorbid with several medical and psychiatric disorders, but has not been tested in HF. The purpose of this exploratory developmental research is to test the feasibility, acceptability, and size of the effects of CBT-I on subjective and objective characteristics of sleep and insomnia symptoms and functional performance in patients with stable HF. Forty patients with stable HF will be randomized to 7 weeks of CBT-I or 7-weeks of HF self-management education with sleep hygiene (attention control). Subjective (diaries, questionnaires) and objective (wrist actigraphy) characteristics of sleep; symptoms, and self-reported functional performance will be measured pre- and post-intervention. The investigators will also obtain day and night measures of urinary free cortisol, free epinephrine/norepinephrine, and melatonin sulfate. They will: 1) refine the protocol, procedures, patient materials, and training manual for the CBT-I intervention and a group HF self-management class (attention-control); 2) evaluate the feasibility and acceptability of the CBT-I intervention and the attention-control conditions; 3) evaluate the size of the effects of group CBT-I, compared with attention-control, on objective (actigraph) and subjective (questionnaire and sleep diary) sleep characteristics, self-report of insomnia symptoms, and beliefs and attitudes about sleep; and 4) evaluate the size of the effects of CBT-I, compared with attention-control, on daytime symptoms (fatigue, depression, anxiety, excessive daytime sleepiness) and functional performance. The primary outcome will be self-reported sleep continuity (sleep efficiency). Investigators will also explore the effects of changes in characteristics of sleep and insomnia symptoms on symptoms and daytime function; the effects of CBT-I, compared with attention control, on nocturnal symptoms, and the effects of CBT-I, compared with attention control, on biological indicators of nocturnal and daytime Hypothalamic Adrenal Pituitary axis (urinary free cortisol), sympathetic nervous system (urinary epinephrine/norepinephrine, and pineal (urinary melatonin) function. The results will be used to support design decisions for a future larger scale efficacy study and may ultimately lead to translation of CBT-I into the care of patients with HF.

ELIGIBILITY:
Inclusion Criteria:

* Stable chronic heart failure
* reports of difficulty initiating or maintaining sleep or waking too early in the morning
* English speaking/reading

Exclusion Criteria:

* untreated sleep disordered breathing or restless legs syndrome
* rotating/night shift work
* active illicit drug use
* bipolar disorder
* neuromuscular conditions affecting the non-dominant arm
* end-stage renal failure
* significant cognitive impairment
* unstable medical or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Insomnia severity | baseline two weeks after completing treatment or attention/control
  Insomnia severity will be measured with the Insomnia Severity Index, a brief self-report instrument measuring patients' perception of their insomnia. The instrument includes 7 items assessing the severity of sleep onset and sleep maintenance difficulties, satisfaction with current sleep pattern, interference with daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Each item is rated on a 0-4 scale (4 indicates greater severity) with a total score ranging from 0 to 28. Scores are categorized as not clinically significant, subthreshold insomnia, moderate insomnia or severe insomnia.

SECONDARY OUTCOMES:
Depressive symptoms | Baseline and two weeks after completing treatment or attention control
  Depressive symptoms will be measured with the Center for Epidemiological Studies Depression Scale, a 20 item self-report instrument used to measure symptoms of depression in nine different groups as defined by the American Psychiatric Association Diagnostic and Statistical Manual, fifth edition. These symptom groups include sadness, loss of Interest, appetite, sleep, thinking/concentration, guilt, fatigue, agitation, and suicidal ideation. Possible scores range from 0-60, and determination of depressive symptom category (no clinical significance, subthreshhold depression symptoms, possible major depressive episode, probable major depressive episode, and meets criteria for major depressive episode) is based upon an algorithm.
Sleepiness | Baseline and two weeks after completing treatment or attention control
  Sleepiness will be measured using the Epworth Sleepiness Scale (ESS) a report instrument used to measure general levels of daytime sleepiness or sleep propensity in adults. The instrument asks subjects to rate on a scale of 0 to 3 the chances that he or she would doze in each of eight different situations. ESS scores can range from 0 to 24, with higher scores indicating higher levels of daytime sleepiness.
Anxiety | Baseline and two weeks after completing treatment or attention-control
  Anxiety will be measured with the Spielberger State Anxiety Inventory (STAI), a self-report instrument to measure the presence and severity of current symptoms of anxiety. The instrument includes 20 items to evaluate the current state of anxiety, using items that measure subjective feelings of apprehension, tension, nervousness, worry, and activation/arousal of the autonomic nervous system. Scores range from 20-80, with higher scores indicating greater anxiety.
Fatigue | baseline and two weeks after completing treatment or attention-control
  The symptom of fatigue will be measured with the Multidimensional Assessment of Fatigue Scale, a 16 item self-report instrument that measures fatigue according to four dimensions: degree and severity, distress that it causes, timing of fatigue, and its impact on various activities of daily living. The items are used to calculate scores for each of the four dimensions listed, as well as a global fatigue index (GFI). A higher score indicates more severe fatigue, fatigue distress, or impact on activities of daily living.
Sleep efficiency | baseline and two weeks after completing treatment or attention control
  Sleep efficiency refers the ratio of time spent asleep to the amount of time spent in bed. Sleep efficiency will be subjectively measured with the Pittsburgh Sleep Quality Index, an instrument used to calculate self-reported sleep duration, sleep efficiency sleep latency, sleep disturbances, and global sleep quality. The 19 self-rated items are calculated to provide a global score ranging from 0-21, with "0" indicating no difficulty, and "21" indicating severe difficulty in all areas. Sleep efficiency will also be objectively measured using actigraphy, a method of inferring sleep from the presence or absence of wrist movement. Participants will wear the Respironics Minimitter Actiwatch AW2, a wrist-worn actigraph, to elicit objective sleep efficiency for a two week period. Participants will also complete a daily diary (lights out/on, times/purpose of removal, hypnotic use) for use in interpretation of actigraphy data.
Functional Performance | baseline and two weeks after completing treatment or attention control
  Functional performance will be measured with the Medical Outcomes Study (MOS) SF36v2 Physical Functioning Scale. The SF36v2 is a multi-purpose self-reported health survey that yields an 8-scale profile of functional health and well-being. The physical functioning scale assesses performance of daily activities, with the lowest score indicating an individual who is very limited in performing all physical activities, including bathing or dressing, and the highest score indicating an individual who can perform all types of vigorous physical activity without limitations due to health.
Thoughts and beliefs about sleep | Baseline and two weeks after completing treatment or attention control.
  This will be measured with a 16 item likert scale. The Dysfunctional Beliefs and Attitudes about Sleep Scale
Cortisol | baseline and two weeks after completing treatment or attention control.
  We will measure urinary free cortisol as a biological measure of stress. Participants will provide urine specimens in the morning (from the previous night) and again late in the afternoon (reflecting the afternoon). This will enable understanding of both day and night levels of stress.
Melatonin | baseline and two weeks after completing treatment or attention control.
  We will measure melatonin as a biological measure of the circadian rhythm. Participants will provide urine specimens in the morning (from the previous night) and again late in the afternoon (reflecting the afternoon). This will enable understanding of both day and night levels of stress.
Epinephrine | baseline and two weeks after completing treatment or attention control.
  We will measure epinephrine ("adrenaline") as a biological measure of stress. Participants will provide urine specimens in the morning (from the previous night) and again late in the afternoon (reflecting the afternoon). This will enable understanding of both day and night levels of stress.
Norepinephrine | baseline and two weeks after completing treatment or attention control.
  We will measure norepinephrine as a biological measure of stress. Participants will provide urine specimens in the morning (from the previous night) and again late in the afternoon (reflecting the afternoon). This will enable understanding of both day and night levels of stress.
Nocturnal symptoms | baseline and two weeks after completing treatment or attention control
  We will measure shortness of breath, nocturnia, and pain. Participants will complete a daily diary each morning upon awakening and indicate on a 10 item numeric scale the degree to which they experienced these symptoms during the past night.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy S. Redeker, PhD, RN, Principal Investigator — Yale University School of Nursing
Locations (1):
- Yale University School of Nursing, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Redeker NS, Jeon S, Andrews L, Cline J, Jacoby D, Mohsenin V. Feasibility and Efficacy of a Self-Management Intervention for Insomnia in Stable Heart Failure. J Clin Sleep Med. 2015 Oct 15;11(10):1109-19. doi: 10.5664/jcsm.5082. PMID 25979100
- [Derived] Breazeale S, Jeon S, Hwang Y, O'Connell M, Nwanaji-Enwerem U, Linsky S, Yaggi HK, Jacoby DL, Conley S, Redeker NS. Sleep Characteristics, Mood, Somatic Symptoms, and Self-Care Among People With Heart Failure and Insomnia. Nurs Res. 2022 May-Jun 01;71(3):189-199. doi: 10.1097/NNR.0000000000000585. PMID 35149627
- [Derived] Redeker NS, Jeon S, Andrews L, Cline J, Mohsenin V, Jacoby D. Effects of Cognitive Behavioral Therapy for Insomnia on Sleep-Related Cognitions Among Patients With Stable Heart Failure. Behav Sleep Med. 2019 May-Jun;17(3):342-354. doi: 10.1080/15402002.2017.1357120. Epub 2017 Aug 22. PMID 28745520